CLINICAL TRIAL: NCT07155382
Title: Allogeneic Hematopoietic Cell Transplantation From Donor- Sources of Matched-sibling, Matched-unrelated, or Haploidentical- Family Donors Using Uniform Conditioning Regimen of Busulfan, Fludarabine, and Antithymocyte Globulin for Acute Myeloid Leukemia in Remission - an Observational Study
Brief Title: Allogeneic HCT Using Conditioning Regimen of BuFluATG for AML CR1
Status: Completed | Type: Observational
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Yunsuk Choi, Associate professor, Asan Medical Center
Other Study IDs: Allogeneic HCT for AML CR1
Record Dates: First submitted 2025-08-25; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Allogeneic HCT for AML CR1
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
1. Study Objectives

   * To evaluate the effect of various clinical variables including HLA-disparity and NK cell-related variables, upon outcomes of allogeneic hematopoietic cell transplantation (HCT) using uniform conditioning regimen including busulfan, fludarabine, and antithymocyte globulin (ATG) in patients with acute myeloid leukemia (AML) in the first complete remission (CR). The donors for allogeneic HCT include HLA-matched siblings, matched unrelated donors, and haploidentical family donors.
   * The endpoints of the study are engraftment, secondary graft failure, acute and chronic graft- versus-host disease (GVHD), immune recovery, infections, leukemia recurrence, non-relapse mortality, and relapse-free (RFS) and overall survival (OS) of patients.
2. Patient Eligibility

   * Patients with non-promyelocytic AML (intermediate-risk or high-risk diseases by NCCN guideline 2016) in the first CR
   * Patients should be 16 years of age or more and 75 years of age or less
   * The performance status of the patients should be 70 or over by Karnofsky performance scale
   * Patients should have adequate hepatic function (bilirubin less than 2.0 mg/dl, AST less than three times the upper normal limit)
   * Patients should have adequate renal function (creatinine less than 2.0 mg/dl)
   * Patients should have adequate cardiac function (ejection fraction > 40% on MUGA scan)
   * Patients and stem cell donors must sign informed consent
   * For hematopoietic cell donor, if a patient has an HLA-matched sibling (65 years or younger), that sibling will be a cell donor. If a patient does not have an HLA-matched sibling but an HLA-A, B, C, DRB1 7-8/8 matched unrelated donor, the unrelated donor will be a cell donor. If a patient has neither HLA-matched sibling nor unrelated donor, an HLA-haploidentical familial donor will be a cell donor.
3. Treatment Plan

   Patients in the study will receive conditioning therapy with busulfan, fludarabine, and antithymocyte globulin. If patients are 54 years old or younger, the patients will receive three days' busulfan administration. If patients are older than 54 years or have co-morbidity, the patients will receive two days' busulfan administration. Graft is non-T cell depleted mobilized peripheral blood hematopoietic cells. GVHD prophylaxis will be given with cyclosporine 1.5 mg/kg iv infusion q12 hrs beginning day -1; methotrexate 15 mg/m2 iv push one day after HCT, then 10 mg/m2 3 days and 6 days after HCT
4. Treatment Evaluation

Regimen related toxicities will be graded by NCI, Common Toxicity Criteria, v 4.0. The status of mixed chimerism will be evaluated by PCR analysis of short tandem repeats (STRs) of one of nine polymorphic introns or amelogenin. The chimerism status will be analyzed from mononuclear cells on 1, 3, and 6 months after HCT. Immune recovery of the patients after stem cell transplantation will be monitored by lymphocyte subset count and measurement of Ig G, Ig M, Ig A levels and Ig G subset (G1, G2, G3) on 1, 3, 6, and 12 months. In the study, at least 200 evaluable cases of HCT will be performed.

DETAILED DESCRIPTION:
1.0 STUDY OBJECTIVES

To evaluate the effect of various clinical variables including HLA-disparity and NK cell-related variables upon outcomes of allogeneic hematopoietic cell transplantation (HCT) in patients with acute myeloid leukemia (AML) in the first complete remission (CR). The donors for allogeneic HCT include HLA-matched siblings, matched unrelated donors, and haploidentical family donors. Uniform conditioning regimen of busulfan, fludarabine, and antithymocyte globulin (ATG) will be used regardless of donor-sources.

The endpoints of the study are engraftment, secondary graft failure, acute and chronic graft- versus-host disease (GVHD), immune recovery, infections, leukemia recurrence, non-relapse mortality, and relapse-free (RFS) and overall survival (OS) of patients.

2.0 BACKGROUND INFORMATION

2.1. Allogeneic HCT is now considered the standard treatment procedure for patients with intermediate- or high-risk AML who achieve CR after induction chemotherapy. Numerous factors have been described to affect allogeneic HCT outcomes and include patient age, performance status, disease risk, HCT methodology (conditioning therapy, GVHD prophylaxis), graft (bone marrow vs. peripheral blood mononuclear cells, cell dose), donor-patient HLA- disparity, and donor-patient natural killer cell alloreactivity. Of those, HLA-disparity was considered the most important determinant of HCT outcomes and, therefore, traditionally, allogeneic HCT was performed from HLA-matched sibling (MSD) or unrelated donors (MUD). Recent innovations in HCT mothodologies, such as reduced-intensity conditioning (RIC), anti- thymocyte globulin (ATG) in conditioning regimen, and post-transplantation cyclophosphamide made HCT from HLA-haploidentical family donors (HFD) feasible. In fact, HFD-HCT using aforementioned approaches resulted in consistent donor cell engraftment and low rates of acute and chronic GVHD and non-relapse mortality (NRM). Currently, in many institutions including ours, HFD-HCT is performed as a part of routine clinical practice for patients with AML in remission when they have no HLA-matched sibling or unrelated donor available. Successful HCT from HFD showed that HLA-haplotype barrier between the donor and patient, i.e., 3-4 mismatches/8 HLA-A, -B, -C, and DR antigen can be overcome for successful allogeneic HCT, which contradicts the traditional concept of allogeneic HCT, whereby >1 antigen mismatch was considered the most important cause for increased graft failure, increased acute and chronic GVHD, delayed immune reconstitution, and NRM. Incorporation of ATG in the conditioning regimen is probably one of major factors that attenuated HLA-disparity effect in HFD-HCT. In unrelated donor HCT, HLA-mismatch between donor and patient was not a significant determinant for HCT outcomes when ATG was used in conditioning regimen. Furthermore, GVHD-modulating effect of ATG was well- documented in a randomized trial of unrelated donor-HCT using myeloablative conditioning, where the inclusion of ATG-Fresenius 20 mg/kg/day 1-3 days before donor cell transplantation was shown to decrease grade III-IV acute GVHD (24.5% to 11.7%; P=0.054) and extensive chronic GVHD (42.6% to 12.2%; P<0.0001). Likewise, in a randomized trial of MS-HCT using myeloablative conditioning and peripheral blood grafting, inclusion of ATG-Fresenius 10 mg/kg/day 1-3 days before transplantation resulted in decrease in grade II-IV acute GVHD (18.1% to 10.8%; P=0.13) and chronic GVHD (68.7% to 32.2%; P<0.001). In our phase 2 study of allogeneic HCT in AML in remission, patients undergoing MU- and HF-HCT received same RIC containing busulfan, fludarabine, and ATG (Thymoglobulin, 9 mg/kg), while patients undergoing MS-HCT received myeloablative busulfan-cyclophosphamide conditioning (71%) or RIC containing lower dose of ATG (29%; Thymoglobulin 4.5 mg/kg). Surprisingly, the 2-year cumulative incidence of moderate-to-severe chronic GVHD higher for MS-HCT (40%) that for MUD- or HFD-HCT (both 22%; P=0.02), which suggested that ATG in the conditioning rather than HLA-disparity is stronger determinant for chronic GVHD occurrence . These data showed that ATG added to the conditioning regimen can decrease GVHD, especially chronic GVHD, in HLA-mismatched, as well as matched-donor HCT settings. A Japanese registry study showed that the significance of HLA-allele mismatch in terms of grade III-IV acute GVHD and survival in unrelated donor HCT changed over the years with less impact in recent cohort of patients (after 2002) than in previous cohort of patients (before 2002).

2.2. Other clinical variables that have been shown to affect HCT outcomes in AML are those related to natural killer (NK) cell alloreactivity. Lack of HLA ligand for donor inhibitory killer immunoglobulin-like receptors (KIR) was correlated with decreased recurrence in AML, but not in acute lymphoblastic leukemia (ALL), after HLA-matched sibling or unrelated donor HCT. Furthermore, in terms of donor KIR genotype, presence of KIR B/x-haplotype, when compared to A/A-haplotype, was associated with better RFS and OS in unrelated-donor HCT. Presence of activating donor KIR2DS1 in association with type 2 HLA-C was shown to be associated with decreased AML relapse after unrelated donor HCT. Polymorphism in donor KIR2DL1 was shown to be correlated to AML and ALL leukemia progression and patient survival. In a study of donor NK cell infusion after HFD-HCT in refractory acute leukemia, stronger expression of activating receptors, particularly NKp30, was shown to be correlated with CR and less leukemia recurrence after HCT. There are reports, however, showing contradicting data regarding association between donor KIR phenotyping and HCT outcomes. Furthermore, these studies investigating prognostic effect of NK cell-related variables are either retrospective or post-hoc analysis and, therefore, need to be confirmed in prospective studies.

2.3. To ascertain the significance of HLA-disparity or NK cell related variables affecting HCT outcomes, they need to be evaluated in a prospective study setting. Furthermore, use of uniform method of transplantation procedure in a patient cohort with single disease entity would be preferred. Successful advent of HFD-HCT using ATG in conditioning regimen made allogeneic HCT feasible after the same conditioning regimen regardless HCT donors of MSD, MUD, and HFD. In our current study, patients with AML in the first CR status will be treated with allogeneic HCT using uniform conditioning regimen of busulfan (dose adjusted for patients' age), fludarabine, and ATG. Furthermore, mobilized peripheral blood mononuclear cells, which are used increasingly in matched as well as in mismatched HCT settings, rather than bone marrow cells will be used as graft. In this prospective cohort of patients, various clinical variables, including HLA-disparity, HCT donor-type, and NK cell related variables will be evaluated for their prognostic significance.

3.0 PATIENT ELIGIBILITY

3.1. Patients with non-promyelocytic AML, intermediate- or poor-risk categories by NCCN ver 2 (2016) guidelines , who achieve CR after induction chemotherapy.

3.2. Patients should be 16 years of age or more, and 75 years of age or less. 3.4. The performance status of the patients should be 70 or over by Karnofsky performance scale.

3.5. Patients should have adequate hepatic function (bilirubin less than 2.0 mg/dl, AST less than three times the upper normal limit).

3.6. Patients must have adequate renal function (creatinine less than 2.0 mg/dl).

3.7. Patients must have adequate cardiac function (ejection fraction > 40% on MUGA scan).

3.8. Patients must sign informed consent.

Donor selection process

3.9. Donor selection process may begin before or when the patients achieve CR. 3.9.1. If a patient has a willing HLA-matched sibling of 65 years or younger, that sibling will be a cell donor.

3.9.2. If a patient has no HLA-matched sibling of 65 years or younger, but a willing HLA- matched unrelated donor is available (younger than 55 years as regulated by KMDP), this will be a cell donor. The donor must be matched with the patient for 7-8 of 8 HLA-A, -B, -C, and -DRB1 allele match.

3.9.3. If a patient does not have an HLA-matched sibling nor unrelated donor, but an HLA- haplotype mismatched family member (offspring, parents, haploidentical sibling) available, this will be a cell donor.

3.9.4. Hematopoietic cell donor must sign informed consent.

4.0 TREATMENT PLAN

4.1. All patients will be registered to the BMT coordinator, Young-Shin Lee, RN, CNS or Mijin Jeon, RN, CNS.

4.2. The patients will have a triple-lumen Hickman central-venous catheter (CVC) placed. Chest X-ray should be taken after CVC placement to confirm the location of CVC and absence of hematoma formation or pneumothorax.

4.3. Lumbar puncture will be done and intrathecal preservative free methotrexate 15 mg will be given.

4.4. Menstruating women will be given gonadotrophin-release hormone agonist or Provera 10 mg po daily.

4.5. The preparative regimen (Bu-Flu-ATG) 4.5.1. Busulfan (Bu) 3.2 mg/kg/day iv daily on days -7, -6, and -5. Patients who are ≥55 years of age or with co-morbidity will receive Bu for 2 days only (days -7 and -6).

4.5.2. Fludarabine (Flu) 30 mg/m2/day in D5W 100 ml iv over 30 minutes starting at 4 pm daily on days -7, -6, -5, -4, -3, and -2.

4.5.3. Methylprednisolone 2 mg/kg in D5W 100 ml iv over 30 minutes on days -4, -3, -2, and -1.

4.5.4. Anti-thymocyte globulin (ATG, Thymoglobulin, Genzyme Transplant, Cambridge, MA, USA) 3.0 mg/kg/day (for haploidential family or unrelated donor) or 1.5mg/kg/day (for matched sibling donor) in N/S 500-800 ml (less than 4 mg/ml) iv over 4 hours starting at 8 am daily on days , -3,-2 and -1.

4.6. Hematopoietic stem cell collection from the donors 4.6.1. Recombinant human granulocyte colony-stimulating factor (G-CSF, Filgrastim) 10 mcg/kg will be administered sc to stem cell donors daily for 4 days (from day -3 to day 0).

4.6.2. Daily CBC will be done. 4.6.3. Starting day 4 of G-CSF administration (day 0), peripheral blood mononuclear cells will be collected by leukapheresis for 1-2 days (days 0; or 0 and 1). A sample will be taken for cell count of total nucleated cells, CD34+ cells, CD3+ cells, CD4+ cells, CD8+ cells, and CD56+ cells.

4.6.4. After the sampling, the final product collected on day 0 and 1 will be infused to the patients immediately on day 0 and day1, respectively.

4.6.5. At least 3x106/kg of CD34+ cells should be collected on day 0. If not, additional collection may be scheduled under the discretion of attending physician.

4.7. Peripheral blood hematopoietic cell infusion (day 0; or days 0-1). 4.7.1. For ABO matched or minor mismatched transplantation, premedication with chlorpheniramine 4 mg iv push and acetaminophen 600 mg po will be given. Stem cells will be infused via CVC over 1 hour.

4.7.2. For major ABO mismatched transplantation, premedication with chlorpheniramine 4 mg iv push, acetaminophen 600 mg po, 10% mannitol 100 g iv over 4 hours beginning 30 minutes before stem cell infusion, and hydrocortisone 250 mg iv immediately before and 30 minutes of stem cell infusion will be given. Stem cells will be infused via CVC over 1 hour.

4.8. Supportive cares. 4.8.1. Dilantin 15 mg/kg (ABW) in NS 200 ml iv over 1 hour for loading on day -8, then 200 mg po bid through -5.

4.8.2. Clotrimazole powder to groin, axilla, and perianal area bid from day -8 until absolute neutrophil count (ANC) > 3,000/㎕.

4.8.3. Sodium bicarbonate/saline mouthwash qid until mucositis is resolved. 4.8.4. Micafungin 50 mg iv qd from Day 1 to ANC > 3,000/㎕. 4.8.5. Ciprofloxacin 500 mg po bid (for selective bowel decontamination) until ANC > 3,000/㎕. With the first fever spike, ciprofloxacin is discontinued and broad spectrum antibiotics are begun.

4.8.6. Acyclovir 250mg/ m2 iv twice a day will be given from day 1, and will be changed into acyclovir 400mg po bid until the discontinuation of cyclosporine administration.

4.8.7. Letermovir 240 mg po or IV until D100 in patients with positive CMV IgG and negative CMV PCR after PBSC infusion. Discontinue if CMV PCR is positive.

4.8.8. The patients are hydrated with 0.9 % NS at 100 ml/hr while the patients are receiving busulfan.

4.8.9. rhG-CSF (Grasin) 450 ㎍ in 100 ml of D5W will be given iv over 3 hours daily from day 5 until ANC>3,000/㎕.

4.8.10. Bactrim 2 t po qd three times a week when ANC>3,000/㎕. 4.8.11. Intravenous immunoglobulin 500 mg/kg (ABW) iv over 6 hours q o week starting day 7 until day 90 then q month until day 180.

4.9. GVHD prophylaxis 4.9.1. Cyclosporine 1.5 mg/kg in N/S 100 ml iv over 2-4 hours q12 hrs beginning day -1. Adjust cyclosporine dose to provide appropriate blood level and according to the change of renal function.

4.9.2. Methotrexate 15 mg/m2 iv on one day, 10mg/m2 iv on 3 days, and 6 days after the last day of donor cell infusion.

4.9.3. Cyclosporine dosing will be changed to oral dosing when oral feeding became feasible at the twice the i.v. dosages. Provided that there is no GVHD, cyclosporine dose will be tapered by 10% every 2-4 weeks starting day 30 of HCT.

4.10. Cytomegalovirus (CMV) prophylaxis and Epstein-Barr virus (EBV) monitoring 4.10.1. Blood CMV quantitative PCR will be done weekly and EBV quantitative PCR will be done biweekly (once per two weeks) starting day -7 until day 100. CMV prophylaxis with ganciclovir will be considered when peripheral blood ANC is over 3,000/mcl and CMV quantitative PCR is positive; ganciclovir 5 mg/kg iv (every 12 hours for 7 days then) once daily until 1-2 weeks after the negative conversion of CMV quantitative PCR.

4.11. CNS prophylaxis: Intrathecal methotrexate administration will be resumed after the patient recovered platelet count to over 50,000/mcl. Methotrexate 15 mg will be given intrathecally once every 2 weeks for three times (total four doses including one given before preparatory regimen).

5.0 TREATMENT EVALUATION

5.1. Donor work up will include;

* HLA-A, -B, -C, and -DR typing based on serologic typing (for sibling matched donor) or based on PCR-sequencing methods(for unrelated donor or mismatched familial donor), ABO/Rh typing, CBC with reticulocyte count, chemistry, BUN/phosphorus, electrolytes, coagulation battery, urinalysis with microscopy, EKG, chest PA and lateral, HBsAg, HBsAb, HCV Ab, HIV Ab, VDRL, CMV(Ig G), HSV(Ig G), EBV serology, Toxoplasma titer (Ig G), VZV (Ig G).
* Immunophenotyping of lymphocytes using 6-color flow cytometry
* Analysis of gene expression according to lymphocytes subset using RNA sequencing

5.2. Patient work up will include;

* HLA-A, -B, -C, and -DR typing based on PCR-sequencing methods, ABO/Rh typing, CBC with reticulocyte count, chemistry, BUN/phosphorus, electrolytes, coagulation battery, urinalysis with microscopy, MUGA scan or echocardiogram, dental consult and Panorex films, ENT consult and PNS films, PFT with DLCO, Urinalysis, Chest X-ray, EKG, diagnostic LP with fluid battery (cell count, glucose, protein, LD, fungal and bacterial cultures, cytospin), bone marrow aspirate and biopsy with cytogenetics and appropriate molecular tests such as bcr-abl, aml1-eto, HBsAg, HBsAb, HBcAb (IgG), HCV Ab, HIV Ab, VDRL, CMV (IgG, IgM), HSV (IgG, IgM), EBV serology, Toxo titer (IgG), VZV (IgG), ABGA, serum pregnancy test ((beta-hCG) ) in females, CBC with reticulocyte, chemical batt with BUN/P, coagulation batt with fibrinogen, ABO and Rh type, blood CMV antigenemia and quantitative CMV and EBV PCR, and isoagglutinin titers if ABO mismatched BMT.
* Immunophenotyping of lymphocytes using 6-color flow cytometry
* Analysis of gene expression according to lymphocytes subset using RNA sequencing

5.3. The diagnosis of GVHD will be made according to the criteria in Appendix VI. The diagnosis of hepatic veno-occlusive disease of the liver (VOD) will be made according to the criteria of McDonald et al. RRT will be graded by NCI, Common Toxicity Criteria v3.0.

5.4. The status of mixed chimerism will be evaluated by PCR analysis of short tandem repeats (STRs) of one of nine polymorphic introns or amelogenin. The chimerism status will be analyzed from mononuclear cells on 1, 3, 6 months after HCT.

5.5. Immune reconstitution including absolute numbers, immunophenotyping, and gene expression changes will be analyzed at 2 weeks, 4 weeks, and 3 months, 6 months, and 12 months after HCT. If acute or chronic GVHD develops, additional blood sample will be obtained for immune cell analysis. If skin or endoscopic biopsy is performed to confirm the GVHD diagnosis, additional tissue samples will also be obtained simultaneously.

5.6. Blood CMV quantitative PCR will be done weekly and EBV quantitative PCR assays will be done biweekly (once per two weeks) until day 100 of stem cell transplantation.

5.7. Immune recovery of the patients after stem cell transplantation will be monitored by lymphocyte subset count and measurement of Ig G, Ig M, Ig A levels and Ig G subset (G1, G2, G3) on 1, 3, 6 months after HCT.

5.8. The patients will be followed with physical examination and appropriate blood test including CBC at least every 3 months for 1years after transplantation

ELIGIBILITY:
Inclusion Criteria:

3.1. Patients with non-promyelocytic AML, intermediate- or poor-risk categories by NCCN ver 2 (2016) guidelines (Appendix I), who achieve CR after induction chemotherapy.

3.2. Patients should be 16 years of age or more, and 75 years of age or less. 3.4. The performance status of the patients should be 70 or over by Karnofsky performance scale (Appendix II).

3.5. Patients should have adequate hepatic function (bilirubin less than 2.0 mg/dl, AST less than three times the upper normal limit).

3.6. Patients must have adequate renal function (creatinine less than 2.0 mg/dl).

3.7. Patients must have adequate cardiac function (ejection fraction > 40% on MUGA scan).

3.8. Patients must sign informed consent.

Donor selection process (See appendix III)

3.9. Donor selection process may begin before or when the patients achieve CR. 3.9.1. If a patient has a willing HLA-matched sibling of 65 years or younger, that sibling will be a cell donor.

3.9.2. If a patient has no HLA-matched sibling of 65 years or younger, but a willing HLA- matched unrelated donor is available (younger than 55 years as regulated by KMDP), this will be a cell donor. The donor must be matched with the patient for 7-8 of 8 HLA-A, -B, -C, and -DRB1 allele match.

3.9.3. If a patient does not have an HLA-matched sibling nor unrelated donor, but an HLA- haplotype mismatched family member (offspring, parents, haploidentical sibling) available, this will be a cell donor.

3.9.4. Hematopoietic cell donor must sign informed consent.

Exclusion Criteria:

Patients who do not meet the inclusion criteria

-

Ages: 16 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: Patients with acute myeloid leukemia undergoing allogeneic hematopoietic stem cell transplantation in first remission
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2024-05-27 (Actual); Study Completion 2024-08-22 (Actual)

PRIMARY OUTCOMES:
To evaluate the effect of various clinical variables upon outcomes of allogeneic hematopoietic cell transplantation in patients with acute myeloid leukemia in the first complete remission . | Immune reconstitution including absolute numbers, immunophenotyping, and gene expression changes will be analyzed at 2 weeks, 4 weeks, and 3 months, 6 months, and 12 months after HCT.
  engraftment, secondary graft failure, acute and chronic graft- versus-host disease (GVHD), immune recovery, infections, leukemia recurrence, non-relapse mortality, and relapse-free (RFS) and overall survival (OS)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
Undecided